CLINICAL TRIAL: NCT05266001
Title: GM-CSF for Reversal of Immunoparalysis in Pediatric Sepsis-induced MODS
Acronym: GRACE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: While the study's data safety monitoring board did not invoke harm, there was a trend toward a potential safety concern in addition to noting a low probability of efficacy after randomizing 141 subjects, so the study was terminated early.
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mark Hall, Chief, Critical Care Medicine, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GRACE-2
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Sepsis-induced Multiple Organ Dysfunction Syndrome
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled clinical trial of the drug GM-CSF vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GM-CSF (Active Comparator): Intravenous GM-CSF 125 mcg/m2/day x 7 days
  Interventions: Drug: GM-CSF
- Placebo (Placebo Comparator): Intravenous placebo x 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GM-CSF — same as arm/group description
  Arms: GM-CSF
Other: Placebo — same as arm/group description
  Arms: Placebo

SUMMARY:
The GRACE-2 study is a prospective, multi-center, double-blind, randomized controlled trial of the drug GM-CSF vs placebo in children with sepsis-induced multiple organ dysfunction syndrome (MODS) who have immunoparalysis with mild to moderate inflammation.

DETAILED DESCRIPTION:
The GRACE-2 study is a is a prospective, multi-center, double-blind, randomized controlled trial of the drug GM-CSF vs placebo in children with sepsis-induced multiple organ dysfunction syndrome (MODS) who have immunoparalysis with mild to moderate inflammation. Eligible subjects will undergo centralized immunophenotyping on MODS Day 2. Those who are found to have immunoparalysis (a whole blood LPS-induced TNF-alpha production capacity < 200 pg/ml) with mild to moderate inflammation (serum ferritin level < 2000 ng/ml) will be randomized to receive intravenous (IV) GM-CSF at a dose of 125 mcg/m2/day x 7 days or placebo. The primary outcome variable is the cumulative 28-day Pediatric Logistic Organ Dysfunction (PELOD)-2 score. Secondary outcomes include measures of health-related quality of life and function status at 3 months from randomization.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 weeks corrected gestational age to < 18 years; AND
* Admission to the PICU or CICU; AND
* Onset of ≥ 2 new organ dysfunctions within the last 3 calendar days (compared to pre-sepsis baseline) as measured by the modified Proulx criteria; AND
* Documented or suspected infection as the MODS inciting event.

Exclusion Criteria:

* Weight <3kg; OR
* Limitation of care order at the time of screening; OR
* Patients at high likelihood of progression to brain death in opinion of the clinical team; OR
* Moribund condition in which the patient is unlikely to survive the next 48 hours in opinion of the clinical team; OR
* History of myeloid leukemia, myelodysplasia, or autoimmune thrombocytopenia; OR
* Current or prior diagnosis of hemophagocytic lymphohistiocytosis or macrophage activation syndrome; OR
* Peripheral white blood cell count < 1,000 cells/mm3 as the result of myeloablative therapy OR receipt of myeloablative therapy within the previous 14 days; OR
* Known allergy to GM-CSF; OR
* Known pregnancy; OR
* Lactating females; OR
* Receipt of anakinra or GM-CSF within the previous 28 days; OR
* Resolution of MODS by MODS Day 2; OR
* Previous enrollment in the GRACE-2 study.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Cumulative 28-day Pediatric Logistic Organ Dysfunction (PELOD)-2 score | 28 days from randomization
  Cumulative Pediatric Logistic Organ Dysfunction (PELOD)-2 score through 28 days post-randomization. The range of PELOD-2 score for a given day is 0 - 33 with a higher number being worse.

SECONDARY OUTCOMES:
3-month health-related quality of life | 3 months post-randomization
  Change in Pediatric Quality of Life inventory (PedsQL) score from baseline to 3 months post-randomization. The range of PedsQL scores is from 0 - 100, with higher values corresponding to better quality of life.
3-month functional status | 3 months post-randomization
  Change in Functional Status Score from baseline to 3 months post-randomization. The range of possible FSS score for a given subject is 6 - 30 with a higher score indicating worse function.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Benioff Children's Hospital - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California - Davis, Sacramento, California
  - Benioff Children's Hospital - Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mercy Children's Hospital, Kansas City, Missouri
  - Duke University, Durham, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] VanBuren JM, Hall M, Zuppa AF, Mourani PM, Carcillo J, Dean JM, Watt K, Holubkov R. The Design of Nested Adaptive Clinical Trials of Multiple Organ Dysfunction Syndrome Children in a Single Study. Pediatr Crit Care Med. 2023 Dec 1;24(12):e635-e646. doi: 10.1097/PCC.0000000000003332. Epub 2023 Jul 27. PMID 37498156